CLINICAL TRIAL: NCT01497249
Title: Assessing Fermentability of a Dietary Fiber (FCHO) in Healthy Non-obese Men and Women
Brief Title: Assessing Fermentability of a Dietary Fiber
Acronym: FCHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Ingredion Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FCHO 2011-086
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Nutritional Intervention
Keywords: Dietary Fiber; Blood glucose control; Fermentability; Tolerability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo Beverage
  Interventions: Dietary Supplement: Placebo
- A dietary fiber (FCHO) (Active Comparator): 15g/BID
  Interventions: Dietary Supplement: A dietary fiber (FCHO)

INTERVENTIONS:
Dietary Supplement: A dietary fiber (FCHO) — 15 g twice per day in beverage
  Other Names: FCHO
  Arms: A dietary fiber (FCHO)
Dietary Supplement: Placebo — Placebo drink
  Other Names: PCB
  Arms: Placebo

SUMMARY:
The objective of this study is to provide evidence for its fermentability of a dietary fiber and to collect information regarding potential health opportunities for glucose control as well as tolerability when being consumed over 7 days.

DETAILED DESCRIPTION:
This study is designed as a randomized, 2-arm, treatment-controlled, within-subjects, 8-hour postprandial crossover study, utilizing a multiple sampling paradigm to evaluate fermentability and potential health opportunities for glucose control of a dietary fiber (FCHO) in healthy non-obese men and women. The study will include 2 - 8 h assessments following consumption of the FCHO drink or a placebo drink and will follow with a 7 day feeding period to assess tolerability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* BMI between 18.5 and 29.9 kg/m2, inclusive
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal, or hepatic disease
* No diabetes
* No Gastrointestinal issues

Exclusion Criteria:

* Pregnant and/or lactating or planning for pregnancy
* Allergies or intolerances to foods consumed in the study Fasting blood glucose > 125 mg/dL.
* Vegetarian
* Taking over the counter fiber supplements or other supplements that may interfere with the study procedures or endpoints
* Taking actively probiotics or purposely taking/ subscribing to a diet high in prebiotics.
* Taking prescription medications that may interfere with study procedures or endpoints (eg., antibiotics)
* Subjects with unusual dietary habits (e.g. pica)
* Actively losing weight or trying to lose weight (unstable body weight fluctuations of > 5 kg in a 60 day period)
* Excessive exercisers or trained athletes
* Addicted to drugs and/or alcohol
* Medically documented psychiatric or neurological disturbances
* Smokers (past smokers may be allowed if cessation is > 2 years)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2012-09-28 (Actual); Study Completion 2012-09-28 (Actual)

PRIMARY OUTCOMES:
The fermentation action of a dietary fiber (FCHO) provided in a breakfast test meal in relatively healthy non-obese men and women | 8 hours
  FCHO will be incorporated in a breakfast meal and compared to the same meal without the FCHO. Subjects will be served a breakfast meal with FCHO or without FCHO in a randomly assigned sequence on two separate occasions (visit 1 and visit 2) under fasting conditions.
  Hydrogen (H2) from breath will be measured before the breakfast test meal (baseline/fasting) and every hour: at 1hr, 2hr, 3hr, 4hr, 5hr, 6 hr, 7hr, and 8hr.

SECONDARY OUTCOMES:
The changes in postprandial glucose concentrations after consuming test meals with FCHO drink compared to placebo drink | 8 hours
  FCHO will be incorporated in a breakfast meal and compared to the same meal without the FCHO. Subjects will be served a breakfast meal with FCHO or without FCHO in a randomly assigned sequence on two separate occasions (visit 1 and visit 2) under fasting conditions.
  Blood glucose will be measured before (fasting/baseline) and after breakfast test meal intake for 4hrs: 0, 30 min, 60 min, 120 min, and 240 min and then again after the light lunch meal at 30, 60, 90, 120 post lunch.
The tolerability of treatments over 7 days | 7 days
  After the in-lab study day (visit 1 and visit 2), subjects will go home with the test beverage packs to be consumed daily for 7 days. Subjects will maintain diaries to ensure daily consumption and on day 7 will be asked to complete a brief questionnaire related to gastrointestinal experiences during the week. Identical procedures will take place after both study days, except the assigned treatment will differ.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute for Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided